CLINICAL TRIAL: NCT03111407
Title: Evaluation of Zimmer® iASSIST™ vs. Conventional Instrumentation in Total Knee Arthroplasty: Radiographic, Clinical and Economic Outcomes
Brief Title: iAssist vs. Conventional Instrumentation in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer, GmbH (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSE2012-05K
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Avascular Necrosis; Post-traumatic; Arthrosis; Knee Osteoarthritis
Keywords: primary total knee arthroplasty
MeSH Terms: conditions — Osteonecrosis; Osteoarthritis; Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: 2 groups of patients: 1 will have the knee prosthesis implanted with iAssist and the other with conventional instrumentation.
Who Masked: Participant
Masking Description: Study patients will not know if their knee prosthesis will be implanted with iAssist or with conventional instrumentation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iAssist group (Other): patients will have primary total knee arthroplasty with the iAssist. The iAssist Knee System is a computer assisted stereotaxic surgical instrument system to assist the surgeon in the positioning of orthopedic implant system components intra-operatively. It involves surgical instruments and position sensors to determine alignment axes in relation to anatomical landmarks and to precisely position alignment instruments and implant components relative to these axes.
  Interventions: Procedure: total knee arthroplasty
- conventional instrumentation (Other): patients will have primary total knee arthroplasty with the conventional instrumentation.
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty — surgical procedure in which damaged parts of the knee joint are replaced with an implant.

SUMMARY:
The purpose of this prospective study is to evaluate Zimmer® iASSIST™ with respect to radiographic, clinical and economic outcomes and compared to conventional instrumentation in primary total knee arthroplasty (NexGen or Persona knee implants).

DETAILED DESCRIPTION:
The study design is a prospective, multicenter, comparative outcome study. The study requires each site to obtain IRB (Institutional Review Board) approval prior to study enrollment. All potential study subjects will be required to participate in the Informed Consent Process.

All study subjects will undergo preoperative clinical evaluations prior to their total knee arthroplasty. Investigators will collect clinical data for 12 months. Follow-up clinical visits include 3 and 12 months post-operatively.

The primary endpoint of this study is defined as component alignment as determined using long leg X-Rays. The secondary endpoint will be to evaluate the Knee Society Score, EQ-5D (EuroQol-5Dimensions) scoring system, operating room time, blood loss and complications

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female
* Patient needs a primary total knee replacement using the NexGen LPS Flex or Persona knee implant
* Patient is diagnosed with non-inflammatory degenerative joint disease (e.g., osteoarthritis, post-traumatic arthritis, avascular necrosis, etc.)
* Patient is over 18 years old
* Patient is able to:

  * Understand what participation in the study entails and willing to consent (patient or his/her legal guardian) to participate in the study by signing and dating an IRB/EC (ethics committee) approved inform consent form, and
  * Follow surgeon/staff instructions, and
  * Return for all follow-up evaluations, and
  * Able and willing to undergo a preoperative full-leg, standing radiographs and/or CT-scan
* Patient meets an acceptable preoperative medical clearance and is free of or treated for cardiac, pulmonary, hematological or other conditions that would pose excessive operative risk.
* Patient has a presence of varus or valgus deformity of 15 degrees or less.

Exclusion Criteria:

* Patient is currently enrolled in an investigational new drug or device study.
* Patient has an active infection (including septic knee, distant infection, or osteomyelitis).
* Patient has severe hip arthrosis.
* Patient has neurological disorders (including, but not limited to Parkinson's disease).
* Patient has had a prior ipsilateral unicompartmental knee arthroplasty, TKA, knee fusion or patellectomy.
* Patient has hip or knee ankylosis.
* Patient has inflammatory joint disease.
* Patient has rheumatoid knee arthritis.
* Patient has indications of intra- and/or extra-articular deformations that would eliminate or tend to eliminate adequate implant support or prevent the use of an appropriately sized implant, such as polio, history of tibial plateau fracture, etc.
* Patient has any metal within 150 mm of the joint line for the operative-side knee.
* Patient has knee deformities greater than 15 degrees of fixed varus, valgus, or flexion contracture on initial physical examination.
* Female who is pregnant or lactating.
* Patient currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
* Patient has arterial disease or stents that would exclude the use of a tourniquet.
* Patient has insufficient quality or quantity of bone to support the implant due to prior knee surgery (or surgeries), cancer, metabolic bone disease, osteoporosis/osteopenia (diagnosed or treated with medication), active/old/remote infection, etc.
* Patient has a mental condition that may interfere with his/her ability to give an informed consent or interfere with his/her ability or willingness to fulfill the requirements of the study.
* Patient has a condition that would place excessive demands on the implant (e.g., Charcot's joints, muscle deficiencies, multiple joint disabilities, skeletal immaturity, etc.).
* Patient has collateral ligament insufficiency.
* Patient has an immunosuppressive disorder (e.g., AIDS, etc.) that would require cytotoxic drugs, corticosteroids, large dose of irradiation, or antilymphocytic serum.
* Patient has an existing condition that would, in the opinion of the investigator, compromise participation or follow-up in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vivoda, Ass.Direct, Study Director — Zimmer Biomet
Locations (3):
- Spain (2):
  - Hospital El Angel, S.A., Málaga
  - Hospital Unviersitario Son Espases, Palma de Mallorca
- Universitätsklinik Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 75 patients were intended to be enrolled according to the protocol but only 72 were finally enrolled.
Groups:
- iAssist Group: 45 iASSIST cases have been enrolled in 3 sites between April 2014 and August 2017.
- Conventional Instrumentation Group: 27 conventional instrumentation cases have been enrolled in 3 sites between April 2014 and August 2017.
Period: Overall Study
Arm/Group | iAssist Group | Conventional Instrumentation Group
Started | 45 | 27
Completed | 44 | 26
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Conventional Instrumentation Group: 27 conventional cases have been enrolled in 3 sites between April 2014 and August 2017.
- Total: Total of all reporting groups
Arm/Group | iAssist Group | Conventional Instrumentation Group | Total
Number analyzed (Participants) | 45 | 27 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (7.9) | 70.3 (7.4) | 68.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 17 | 47
  Male | 15 | 10 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight kg [Mean (Standard Deviation); unit: kg] | 81.4 (17.2) | 84.3 (13.0) | 82.5 (15.7)
Body Mass Index (BMI) kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (5.5) | 30.7 (4.6) | 30.5 (5.1)
Height cm [Mean (Standard Deviation); unit: cm] | 163.5 (10.6) | 166.0 (9.6) | 164.5 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Component Alignment
Description: Assess the differences in component alignment, measured by the mean of radiographs, between iASSIST™ and conventional instrumentation in primary total knee arthroplasty (TKA) procedures.
Time Frame: 1 year
Population: Available data of enrolled patients were used for analysis.
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | iAssist Group | Conventional Instrumentation Group
Number analyzed (Participants) | 44 | 26
degree | 179 (2.9) | 178 (3.9)
Statistical Analysis 1: Comparison: iAssist Group vs Conventional Instrumentation Group; Hip Knee Angle value 1 year post surgery: Mean+/- SD (N)(Min, Max) 95%C.I (lower, upper) iAssist group: 179.9 +/-2.9 (44) (171, 185.3) Conventional group: 178.9 +/-3.9 (26) (167, 185); Test type: Equivalence — Data analyzed with SAS Enterprise Guided (version 7.15 HF3, SAS lnstitute lnc., Cary, NC). Significance level set with q = 0.05. Continuous data (e.g. age, weight, EQ-5D) were summarized using mean, standard deviation, minimum, median, maximum and number of observations. Comparison between continuous baseline and patient visits were performed using standard statistical tests (e.g., a t-test, Wilcoxon test, or one-way ANOVA (as appropriate) were performed as required to evaluate the difference); p = 0.2342, t-test, 2 sided

2. Secondary Outcome: Knee Society Score Assessment
Description: Assess the differences in Knee Society Score between iASSIST™ and conventional instrumentation in primary TKA procedures. Higher (and better) score value: 100, lower value: 0.
  Score 80-100 = Excellent Score 70-79 = Good Score 60-69 = Fair Score below 60 = Poor
Time Frame: 1 year
Population: Available data of enrolled patients were used for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iAssist Group | Conventional Instrumentation Group
Number analyzed (Participants) | 44 | 26
score on a scale | 74.7 (12.5) | 72.4 (11.6)
Statistical Analysis 1: Comparison: iAssist Group vs Conventional Instrumentation Group; Knee Society Score Assessment 1 year post surgery: Mean+/- SD (N)(Min, Max) 95%C.I (lower, upper) iAssist group: 74.7 +/- 12.5 [44] (30.2, 78.0, 89.5), 95% C.I. (70.9, 78.5) Conventional group: 72.4 +/- 11.6 [26] (45.0, 75.2, 90.1), 95% C.I. (67.7, 77.1); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4427, t-test, 2 sided

3. Secondary Outcome: Knee Society Score Function
Description: Knee Society Score function asses 12 months postoperatively between iASSIST™ and conventional instrumentation in primary TKA procedures. Higher (and better) score value: 100, lower value: 0.
  Score 80-100 = Excellent Score 70-79 = Good Score 60-69 = Fair Score below 60 = Poor
Time Frame: 1 year
Population: Available data of enrolled patients were used for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iAssist Group | Conventional Instrumentation Group
Number analyzed (Participants) | 44 | 27
score on a scale | 80.5 (13.8) | 78.5 (19.1)
Statistical Analysis 1: Comparison: iAssist Group vs Conventional Instrumentation Group; Knee Soceity Score Function 1 year post surgery: Mean+/- SD (N)(Min, Max) 95%C.I (lower, upper) iAssist group: 80.5 +/- 13.8 [44] (55.0, 80.0, 100.0), 95% C.I. (76.2, 84.7) Conventional group: 78.5 +/- 19.1 [26] (40.0, 80.0, 100.0),95% C.I. (70.8, 86.2); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.6154, t-test, 2 sided

4. Secondary Outcome: EQ-5D Questionnaire
Description: Assess the differences in EQ-5D between iASSIST™ and conventional instrumentation in primary TKA procedures at 12 months postoperatively.
  Comparison of the derived EQ-5D scale and health state between the 2 groups. The EQ-5D questionnaire includes five dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  EQ-5D values range from -0.2 to 1 where the negative values correspond to bad health states (states worse than death), and 1.0 corresponds to perfect health.
Time Frame: 1 year
Population: Available data of enrolled patients were used for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iAssist Group | Conventional Instrumentation Group
Number analyzed (Participants) | 29 | 20
score on a scale | 0.8 (0.2) | 0.8 (0.3)
Statistical Analysis 1: Comparison: iAssist Group vs Conventional Instrumentation Group; EQ-5D score 1 year post surgery: Mean+/- SD (N)(Min, Max) 95%C.I (lower, upper) iAssist group: 0.8 +/- 0.2 [29] (0.0, 1.0, 1.0), 95% C.I. (0.7, 0.9) Conventional group: 0.8 +/- 0.3 [20] (0.1, 0.8, 1.0), 95% C.I. (0.7, 0.9); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4549, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The adverse events were collected preoperatively, intraoperatively and postoperatively (at 3 months ±2 weeks and 12 months ±1 month postoperative).
Arm/Group | iAssist Group | Conventional Instrumentation Group
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/45 | 4/27
Other Adverse Events (participants affected / at risk) | 7/45 | 3/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | iAssist Group (N=45) | Conventional Instrumentation Group (N=27)
Poor alignment in tibia component (Surgical and medical procedures) | 1 | 0
Sepsis in bronchial asthma, infection exacerbation (Infections and infestations) | 1 | 0 — treated with antibiotics and cortisone
Implant failure (Surgical and medical procedures) | 0 | 1 — treated by total knee revision.
Pulmonary embolism (Vascular disorders) | 0 | 1 — treated with Anticoagulation
Lump in the neck: metastasis,as well as in the lungs (General disorders) | 0 | 1 — treated by removal and irradiation.
Patella transverse fracture+dislocation of the prosthesis+tibia shaft fracture+infe (Surgical and medical procedures) | 0 | 1 — adverse events occured in the opposite side (left side).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | iAssist Group (N=45) | Conventional Instrumentation Group (N=27)
Allergic reaction after eating nuts (General disorders) | 1 | 0
Allergic reaction unclear cause (itching, dyspnea, rash) (General disorders) | 1 | 0
Radius fracture (Surgical and medical procedures) | 1 | 0 — treated by surgery
Flexion Contracture (General disorders) | 1 | 1
Allergic reaction (Dafalgan) (General disorders) | 1 | 0 — treated by stopping the drugs and giving zavegyl/zantic
Foot fracture (Surgical and medical procedures) | 1 | 0 — treated by surgery 1 year later
Delayed Wound Healing (Surgical and medical procedures) | 1 | 0 — treated by wound revision and surgery
Fall from the bed (Social circumstances) | 1 | 0 — Patient and the knee were ok.
Pain in the calf (deep vein thrombosis) (Vascular disorders) | 0 | 1 — treated with xarelto 10mg/day for 3 month
patient felt on the floor, he wanted to stand up alone (Social circumstances) | 0 | 1
Patient still had a joint effusion 6 months after surgery (Surgical and medical procedures) | 0 | 1 — treated by joint puncture

LIMITATIONS AND CAVEATS:
Since the first follow-up visits were performed according to the standard of care of each site, they did not occur at the same time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT03111407/Prot_SAP_000.pdf